CLINICAL TRIAL: NCT06543602
Title: A Multi-modal Recognition Model and Efficacy Evaluation for Agitation Behavior in Critically Ill Patients Based on Remote -Ultra-sensitive Detection Wave ---A Multi-center, Open-label, Observational Study
Brief Title: the Multi-modal Evaluation of Agitation in Critically Ill Patients Based on Remote Video-Ultra-sensitive Detection Wave
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: People's Hospital of Quzhou (Other); The Second Affiliated Hospital of Jiaxing University (Other); Zhoushan Hospital of Zhejiang (Unknown); Longquan People's Hospital (Unknown); Fuyang District First People's Hospital of Hangzhou (Unknown); The Third Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024 0135
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Critically Ill Patients
Keywords: Critically Ill; agitation; monitoring; remote
MeSH Terms: conditions — Critical Illness; Psychomotor Agitation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group: monitoring by manual way
- multiple-model monitoring group: agitation monitoring by remote video-radar wave
  Interventions: Diagnostic Test: multi-model monitoring and alert

INTERVENTIONS:
Diagnostic Test: multi-model monitoring and alert — All agitated critically illed patients are monitored by manual and multi-model monitoring and alert system
  Groups: multiple-model monitoring group: agitation monitoring by remote video-radar wave

SUMMARY:
The goal of this observational study is to learn about the effectiveness of the multi-modal evaluation for agitation behavior in critically ill patients based on remote video-Ultra-sensitive detection wave.

The main question it aims to answer is: evaluate the effectiveness of multi-modal evaluation monitoring system for agitated critically ill patients Participants already taking multi-modal evaluation monitoring system as part of their regular medical care for agitated critically ill patients will compare their effectiveness for agitation for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients at risk of agitation in the ICU
* Patients with RASS score -2 and above
* ≦ 65 years old, ≧ 18 years old

Exclusion Criteria:

* The affected party refused to participate in this study
* Missing/incomplete information
* Vulnerable groups such as pregnant women, those who lack the capacity for civil conduct and do not have the consent of their legal representatives
* Maxillofacial trauma, burns, tumors, surgery, etc. affect facial expression
* Patients with limb impairment and amputation
* Spinal cord injury, limb movement/sensory limitations
* Patients with pre-existing neurological/psychiatric diseases
* Patients with malignant tumors
* Patients with infectious diseases
* Patients with terminal disease and dying disease
* Abnormal behavior due to head injury or craniocerebral disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: any patients with agitation
Sampling Method: Non-Probability Sample
Enrollment: 580 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
the correct rate for alerting agitated critically ill patients | 10-15 seconds every agitated patients during stay in ICU

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - the second affiliated hospital, Zhejiang University school of medicine, Hangzhou, Zhejiang
  - SAHZU, Hanzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided